CLINICAL TRIAL: NCT00221208
Title: A Home Based Resistance Training Program for Obese Adults With Type 2 Diabetes
Brief Title: Home Based Resistance Training For Type 2 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Alberta (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OHP - 69441
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Diabetes
Keywords: Diabetes; Resistance Training
MeSH Terms: conditions — Diabetes Mellitus | interventions — Resistance Training

INTERVENTIONS:
Behavioral: Resistance Training

SUMMARY:
This study will investigate the biological and psychosocial benefits of a home-based resistance-training program for sedentary, obese adults living with type 2 diabetes.

DETAILED DESCRIPTION:
Obese individuals with type 2 diabetes will be randomly assigned to either an experimental group where they will perform moderate to high intensity resistance training (50-60% 1RM weeks 1-3 and 70-85% 1RM in weeks 4-16) three times per week for 16 weeks or to a non-training control group. All resistance training will be performed at home using a multigym apparatus. A personal trainer (PT) will come to the homes of each participant in the experimental group to make sure that exercises are being performed safely with the correct technique, and at the prescribed intensity. In the first two weeks, the PT will come to all 3 sessions per week. In weeks 3-4 this will be reduced to 2 times per week, in weeks 5-8 the PT will come once per week and in the last 8 weeks once bi-weekly.

ELIGIBILITY:
Inclusion Criteria:

Type 2 Diabetes Overweight and Obese (BMI>28) Living inside of City limits

Exclusion Criteria:

Ischemic heart disease Osteoporosis Musculoskeletal abnormalities Currently performing resistance training

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54
Dates: Start 2005-04; Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
HbA1c
Muscular strength

SECONDARY OUTCOMES:
Fasting blood glucose, insulin, lipid concentrations, C-reactive protein, body composition (DEXA), exercise adherence, behaviour change, psychosocial predictors of resistance training, quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Ron C Plotnikoff, PhD, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada

REFERENCES:
- [Derived] Plotnikoff RC, Eves N, Jung M, Sigal RJ, Padwal R, Karunamuni N. Multicomponent, home-based resistance training for obese adults with type 2 diabetes: a randomized controlled trial. Int J Obes (Lond). 2010 Dec;34(12):1733-41. doi: 10.1038/ijo.2010.109. Epub 2010 Jun 8. PMID 20531348